CLINICAL TRIAL: NCT07020806
Title: [68Ga]Ga DOTA-5G as a Diagnostic Imaging Agent for Metastatic/Advanced Invasive Lobular Breast Cancer (LBC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Dr. Helen K Chew, University of California Davis (Unknown); Dr. Cameron Foster, University of California Davis (Unknown); Society of Nuclear Medicine and Molecular Imaging (Unknown)
Responsible Party: Principal Investigator, Julie L. Sutcliffe, Ph.D, Professor, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2213682
Record Dates: First submitted 2025-05-21; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Lobular Breast Carcinoma
MeSH Terms: conditions — Carcinoma, Lobular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- [68Ga]Ga-DOTA-5G PET/CT imaging (Experimental): Following an injection of up to 5 mCi of [68Ga]Ga DOTA-5G patients will be undergo PET/CT scans.
  Interventions: Drug: [68Ga]Ga DOTA-5G

INTERVENTIONS:
Drug: [68Ga]Ga DOTA-5G — Patients will be injected with up to 5 mCi of [68Ga]Ga DOTA-5G and imaged at 1 and 2 hours post injection.

SUMMARY:
This is a prospective study using [68Ga]Ga DOTA-5G PET/CT imaging in patients diagnosed with metastatic/advanced invasive lobular breast cancer (LBC).

DETAILED DESCRIPTION:
This is a phase I investigator-initiated study that will investigate [68Ga]Ga DOTA-5G in patients with metastatic/advanced invasive LBC. 30 patients diagnosed with LBC will be enrolled over a 24-month period.

We hypothesize that a) [68Ga]Ga DOTA-5G will detect lesions in patients with invasive LBC, b) [68Ga]Ga DOTA-5G will be safe and well tolerated, and that c) [68Ga]Ga DOTA-5G PET/CT is more sensitive than 18F-FDG PET/CT at detecting lesions.

ELIGIBILITY:
Inclusion Criteria:

* (Ability to understand and willingness to sign a written informed consent document.
* Men and women age ≥ 18 yrs
* Confirmed presence of metastatic/advanced invasive lobular breast cancer and measurable disease per RECIST (version 1.1)
* Available archival tumor tissue
* Eastern Cooperative Oncology Group Performance Status ≤ 2
* Hematologic parameters defined as: Absolute neutrophil count (ANC) ≥ 1000 cells/mm3,Platelet count ≥ 100,000/mm3, Hemoglobin ≥ 8 g/dL.
* Blood chemistry levels defined as: AST, ALT, alkaline phosphatase ≤ 5 times upper limit of normal (ULN), Total bilirubin ≤ 2 times ULN, creatinine clearance >60 mL/min.
* Anticipated life expectancy ≥ 3 months
* Able to remain motionless for up to 30-60 minutes per scan.

Exclusion Criteria:

* Pregnant and lactating women
* Prisoners
* Concurrent malignancy of a different histology that could confound imaging interpretation.
* Patients who cannot undergo PET/CT scanning because of weight limits(>350lbs)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
The ability of [68Ga]Ga DOTA-5G PET/CT imaging to detect lesions | 2 hours from time of injection
  To assess the ability of [68Ga]Ga DOTA-5G PET/CT imaging to detect lesions. Following injection of [68Ga]Ga DOTA-5G patients will be imaged at 1 and 2 hours. Regions of interest will be drawn around lesions and standard uptake values (SUV) calculated. Detection of metastasis by [68Ga]Ga DOTA-5G PET/CT imaging, positive vs. negative based on if SUVmax >2-fold above normal brain, bone, lung, or liver of [68Ga]Ga DOTA-5G in at least one lesion assessed by [68Ga]Ga DOTA-5G PET/CT and identified on [18F]-FDG PET/CT diagnostic imaging.
Safety and tolerability of [68Ga]Ga DOTA-5G based on the incidence of adverse events using CTCAE v 5.0 | Up to 7 days from time of injection
  To evaluate the safety and tolerability of [68Ga]Ga DOTA-5G patients will be followed for up to 7 days for AEs using CTCAE v 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Sutcliffe, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No